CLINICAL TRIAL: NCT04490824
Title: Can Inhalation of KELEA Excellerated Water Reduce the Time Required for Covid-19 Infected Individuals to Become Symptom-Free and to Test Negative Using Either the PCR or Antigen Assay
Brief Title: Inhalation of KELEA Excellerated Water in Covid-19 Infected Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Progressive Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: KELEA-1
Record Dates: First submitted 2020-07-27; First posted 2020-07-29 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Covid19
Keywords: Energy Medicine; KELEA; Inhalation
MeSH Terms: conditions — COVID-19; Respiratory Aspiration | interventions — Hydrotherapy

STUDY DESIGN:
Intervention Model Description: Participants will be sequentially assigned to receive KELEA activated or KELEA depleted water
Who Masked: Participant
Masking Description: The participant will not be informed as to whether the item that is first received is KELEA emitting or inactive. If requested an active item will be sent following receipt of the post inhalation results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treated Then Control Water (Active Comparator): This Arm includes half of the total randomly allocated participants in the study. Participants will initially inhale KELEA Excellerated Water for 2 days followed by inhaling water without an elevated level of KELEA for 2 days, with Covid-19 testing and symptom assessments performed at the ends of both of the 2 days periods.
  Interventions: Device: KELEA Excellerated Water; Device: Water Without an Elevated Level of KELEA
- Control Than Treated Water (Placebo Comparator): This Arm includes half of the total randomly allocated participants in the study. Participants will initially inhale water without an elevated level of KELEA for 2 days followed by inhaling KELEA Excellerated water for 2 days, with Covid-19 testing and symptom assessments performed at the ends of both of the 2 days periods.
  Interventions: Device: KELEA Excellerated Water; Device: Water Without an Elevated Level of KELEA

INTERVENTIONS:
Device: KELEA Excellerated Water — Water with increased kinetic activity as assessed by published methods of the PI
  Other Names: KELEA Activated Water
Device: Water Without an Elevated Level of KELEA — Bottled water without an elevated level of KELEA, as shown by proprietary testing will be provided as a control.
  Other Names: Control Water

SUMMARY:
Preliminary reports have been received from several sources that the periodic inhaling of the nebulized mist from water that has a heightened level of kinetic activity has quickly (less than 2 days) lessened the severity of symptoms in Covid-19 infected patients. On at least several occasions, a repeat PCR test performed several after inhaling a particular water-based product was negative. There are no perceived adverse effects from inhaling the water mist by using a nebulizer or humidifier. It is important, however, to validate these preliminary findings and to include the inhaling of the mist from water, which does not have an elevated level of kinetic activity. This will be by performed in a patient-blinded manner by sequentially inhaling the two types of water over consecutive 2-day periods with Covid-19 testing at the end of each of the two day periods. Participants will be randomized as to whether they are to inhale the mist from the test or the control water.

DETAILED DESCRIPTION:
Several producers of activated water have been in frequent communication with the Principal Investigator (PI) over the last decade or longer. They have regularly supplied their water products to the PI for laboratory testing, including measuring an activity attributed to the absorption of an environmental force, referred to by the PI as KELEA, an abbreviation for Kinetic Energy Limiting Electrostatic Attraction. KELEA is regarded as the source of cellular energy for the body's alternative cellular energy (ACE) pathway. This pathway can provide a non-immunological defense mechanism against infections, presumably including coronaviruses. The proposed study is to test water products from several suppliers, as well as a naturally available source of KELEA activated water in symptomatic individuals who have tested positive by either PCR or antigen testing for Covid-19. The mode of administration will be by inhalation using a nebulizer or diffuser. Several deep inhalations will be taken on 5 occasions daily. Prior to the first inhalation and at the end of the second day of inhalation, swabs will be taken for Covid-19 PCR and/or antigen testing. Randomly allocated participants will either blindly first test the KELEA excellerated water for two days, followed by using water without an elevated level of KELEA and vice versa. The severity of symptoms will also be monitored at the end of each of the two-days periods of inhalation.

ELIGIBILITY:
Inclusion Criteria: Individuals entering into quarantine because of a positive Covid-19 test using either PCR or an authorized antigen assay. It is not necessary, but preferable, for the participant to be symptomatic for Covid-19 -

Exclusion Criteria: Unwilling to do repeat PCR and/or antigen testing or to provide the results of the repeat testing or the requested clinical data

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Inhalation of KELEA Excellerated Water in Covid-19 Infected Individuals | Two consecutive 2-days periods of sequential inhalation of test and control water in randomized order followed by Coivid-19 testing at the end of both of the 2-days periods.
  Proportion of Covid-19 Positive Participants Who Subsequently Test Negative Following 2-Days of Inhalation.

SECONDARY OUTCOMES:
Inhalation of KELEA Excellerated Water in Covid-19 Infected Individuals | Two consecutive 2-days periods of sequential inhalation of test and control water in randomized order.
  Proportion of the Symptomatic Participants Who Become Asymptomatic Following 2-Days of Inhalation.

CONTACTS AND LOCATIONS:
Overall Officials: W John Martin, MD, PhD, Principal Investigator — Medical Director
Locations (1):
- Institute of Progressive Medicine, South Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin WJ. Enhancing the Alternative Cellular Energy (ACE) Pathway with KELEA Activated Water as Therapy for Infectious Diseases. Infect Disord Drug Targets. 2021;21(3):314-319. doi: 10.2174/1871526520666200211115111. PMID 32066365